CLINICAL TRIAL: NCT03431597
Title: Effectiveness of a Micronutrient Supplement to Lower Plasma Homocysteine in Non-pregnant Women of Reproductive Age
Brief Title: Effectiveness of a Micronutrient Supplement to Lower Plasma Homocysteine MDEG2 Pilot Supplementation Trial
Acronym: MDEG2-PST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCC 1575
Record Dates: First submitted 2018-01-26; First posted 2018-02-13 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Micronutrient Deficiencies; Hyperhomocysteinemia
MeSH Terms: conditions — Hyperhomocysteinemia

STUDY DESIGN:
Intervention Model Description: 3-arm randomized controlled trial, unblinded, with 125 women per arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oral nutritional supplementation (Experimental): Daily novel micronutrient supplement: 800 μg folic acid, 5.2 μg cyanocobalamin (B12), 2.8 mg Riboflavin-5'- phosphate (B2), 4g trimethylglycine (betaine) in drink powder form. The drink will be dissolved in 200ml of water and taken daily for 12 weeks
  Interventions: Dietary Supplement: novel micronutrient
- oral nutritional supplementation, UNIMMAP (Active Comparator): The United Nations Multiple Micronutrient Preparation (UNIMMAP) supplement is a capsule containing 15 micronutrients (vitamins A, D, E, B1, B2, B6, B12, C, Niacin, Folic Acid, Fe, Zn, Cu, I, Se) at the Recommended Daily Allowance level. UNIMMAP will be provided in capsule form and taken daily with water for 12 weeks.
  Interventions: Dietary Supplement: existing micronutrient supplement, UNIMMAP
- control (No Intervention): no treatment will be given to this group observation only (no placebo)

INTERVENTIONS:
Dietary Supplement: novel micronutrient — The supplements will be supplied to participants on a daily basis. The novel micronutrient supplement will be provided in powder form with instructions to dissolve one sachet in 250ml of clean water
  Arms: oral nutritional supplementation
Dietary Supplement: existing micronutrient supplement, UNIMMAP — UNIMMAP will be provided in tablet form and given one daily
  Arms: oral nutritional supplementation, UNIMMAP

SUMMARY:
This micronutrient supplementation study is a 3-arm randomized controlled trial, unblinded, with 125 women per arm. Non-pregnant, non-lactating healthy women of reproductive age in West Kiang, The Gambia, will be randomized to 12 weeks of daily supplementation of either a) novel micronutrient supplement, b) a United Nations International Multiple Micronutrient Preparation (UNIMMAP) tablet or c) no intervention (control). The novel micronutrient supplement is a drink powder providing 800 µg folic acid, 5.2 µg cyanocobalamin (B12), 2.8 mg Riboflavin-5'-phosphate (B2), and 4g trimethylglycine (betaine). UNIMMAP contains 15 micronutrients at the Recommended Daily Allowance level. The aim is to test the effectiveness of the supplements on correcting micronutrient deficiencies in the dry season and to reduce homocysteine levels. The hypothesis is that the new drink powder will be the most effective supplement, causing a reduction in 1 µmol/L compared to the control group after supplementation.

The supplements will be supplied to participants on a daily basis by Community-based Birth Attendants (CBCs). The CBCs will observe consumption of the supplement. The novel micronutrient supplement will be provided in powder form with instructions to dissolve one sachet in a cup of 200ml water. UNIMMAP will be provided in capsule form to be taken with water. Women will provide one 10ml fasted venous blood sample at baseline and another after 6 and 12 weeks of supplementation. At each time point they will also have their blood pressure and anthropometry assessed and provide a urine pregnancy test.

Correcting micronutrient deficiencies is extremely important for the long-term health of women, and in particular around the time of conception and throughout pregnancy since micronutrients are needed for the proper physical and cognitive development of the baby. Certain micronutrients are required for adding a methyl group to places on DNA ('DNA methylation'). The pattern of these methyl groups can help determine whether a gene is switched on or off. Correct functioning of DNA methylation processes is therefore of critical importance for fetal development. High levels of homocysteine can impede DNA methylation, therefore supplements that reduce homocysteine may not only be beneficial for the mother but also for the developing child. The most effective supplement in this trial will be considered for testing in larger pregnancy trials.

DETAILED DESCRIPTION:
In rural Gambia women experience considerable variation in their diet by season. In the dry season women have particular micronutrient deficiencies that can disrupt one-carbon metabolism pathways. In the dry season women have lower levels of most of the B vitamins and higher levels of homocysteine compared to the rainy season. The goal of this trial is to test two nutritional interventions to see which one works best in providing micronutrients in the ratio and quantity necessary for optimal 1-carbon metabolism in the dry season. The primary end point is to assess which supplement is most effective in reducing plasma homocysteine.

This is a 3-arm randomized controlled trial, unblinded, with 125 women per arm. Non-pregnant, non-lactating healthy women of reproductive age in West Kiang will be randomized to 12 weeks of daily supplementation of either a) novel micronutrient drink powder supplement, b) existing available micronutrient supplement (UNIMMAP) or c) no intervention (control). The novel drink powder provides 800 µg folic acid, 5.2 µg cyanocobalamin (B12), 2.8 mg Riboflavin-5'-phosphate (B2), and 4g trimethylglycine (betaine). This dose is twice the Recommended Daily Allowance for folic acid, B12 and B2. The UNIMMAP tablet provides 15 micronutrients (vitamins A, D, E, B1, B2, B6, B12, C, Niacin, Folic Acid, Iron, Zinc, Copper, Iron, Selenium) at the Recommended Daily Allowance level.

Potentially eligible participants will be identified through the Keneba Health and Demographic Surveillance System in all 35 villages of West Kiang region of The Gambia. Field assistants will visit the homes of potentially eligible participants to provide full information about the purpose and methods of the study, potential risks and benefits, and participants' rights. Full inclusion and exclusion criteria will be assessed. Participants will then be asked to provide a signed or thumb-printed informed consent before being enrolled into the study.

The supplements will be supplied to participants on a daily basis by Community-based Birth Companions (CBCs). The novel drink powder will be provided in daily sachets and dissolved in 200ml water. UNIMMAP will be provided in capsule form to be taken with water. The CBCs will observe consumption of the supplement. Participants will be given 7 coloured cards at the start of each week. Every day they will give the CBC one card and receive their supplement. Each week a field assistant will collect data on compliance by recording card collection in liaison with the CBC.

Women will provide one 10mL fasted venous blood sample at baseline and another after 6 and 12 weeks of supplementation. At each time point they will also have their blood pressure and anthropometry (weight and height) assessed and provide a urine pregnancy test. Women will be brought to the Medical Research Council Gambia (MRCG) field station at Keneba for the baseline, 6 week (mid-line) and 12 week (end-line) data collection visits. Participants will be followed-up after the intervention period for a further 3 weeks to monitor any adverse effects.

The fasted 10mL baseline, 6 week and 12 week blood samples will be taken by venepuncture into EDTA monovettes and kept on ice. Within one hour of collection the samples will be processed by the laboratory in Keneba to centrifuge the samples, separate the plasma and store plasma and red blood cell aliquots at -70°C. One plasma aliquot will be analysed in Keneba to measure homocysteine using the Cobas Integra 400 Plus analyser.

The hypothesis is that the novel micronutrient supplement will reduce plasma by at least 1 µmol/L compared to the control group after 12 weeks of daily supplementation. It will be more effective in reducing plasma homocysteine than existing UNIMMAP tablets.

This trial is powered to study to detect a decrease of 1 µmol/L homocysteine with 80% power and 95% confidence. The trial statistician will use a linear regression model to determine the mean difference between intervention and control homocysteine at 12 weeks adjusted for baseline homocysteine, week 12 age and week 12 body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women aged 18-45 years

  * Non-pregnant, confirmed by pregnancy urine test at eligibility screen
  * Non-lactating (at least 9 months post-partum)
  * No plan to conceive in the ensuing 3 months, asked verbally by field worker
  * No plans to travel
* Healthy with no current illness and no chronic health problems, asked verbally by field worker

Exclusion Criteria:

* Known history of chronic illness (particularly cardiovascular disease, renal disease, thyroid disease, cancer)

  * Taking B vitamin or multivitamin supplements.
  * Taking medication for prevention of seizures (e.g. Carbamazepine).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — A list of eligible women within West Kiang will be generated using the MRCG Keneba Health and Demographic Surveillance System (HDSS) database
Enrollment: 298 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Difference in plasma homocysteine concentration between the drink powder and control arms at end-lineplasma Hcy vs control | after 12 weeks
  To compare the effect of a novel micronutrient supplement taken daily for 12 weeks in the dry season on lowering plasma homocysteine versus the control group supplement taken daily for 12 weeks in the dry season on lowering plasma homocysteine (Hcy) versus the control group

SECONDARY OUTCOMES:
Difference in plasma homocysteine concentration between the drink powder and UNIMMAP arms at end-line | after 12 weeks
  To compare the effect of a novel micronutrient supplement taken daily for 12 weeks in the dry season on lowering plasma homocysteine versus the UNIMMAP group.
Difference in plasma homocysteine concentration between the the drink powder and UNIMMAP arms at mid-line | after 6 weeks
  To compare the effect of a novel micronutrient supplement taken daily for 6 weeks in the dry season on lowering plasma homocysteine versus the UNIMMAP group
Difference in blood pressure (systolic and diastolic) and pulse between the drink powder and control arms at end-line | after 12 weeks
  To compare the effect of a novel micronutrient supplement taken daily for 12 weeks in the dry season on lowering blood pressure and pulse versus the control group

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Prentice, PhD, Principal Investigator — Medical Research Council Unit, The Gambia
Locations (1):
- Keneba Field Station, Banjul, The Gambia

REFERENCES:
- [Derived] James PT, Jawla O, Mohammed NI, Ceesay K, Akemokwe FM, Sonko B, Sise EA, Prentice AM, Silver MJ. A novel nutritional supplement to reduce plasma homocysteine in nonpregnant women: A randomised controlled trial in The Gambia. PLoS Med. 2019 Aug 13;16(8):e1002870. doi: 10.1371/journal.pmed.1002870. eCollection 2019 Aug. PMID 31408467